CLINICAL TRIAL: NCT03379259
Title: Phase 1-2 Study Investigating Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Anti-PD-L1 Monoclonal Antibody BGB-A333 Alone and in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Study of BGB-A333 Alone and in Combination With Tislelizumab in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study Was Terminated Early
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-101; 2018-000265-37 (EudraCT Number)
Record Dates: First submitted 2017-12-11; First posted 2017-12-20 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1A: BGB-A333 monotherapy dose escalation (Experimental)
  Interventions: Drug: BGB-A333
- Phase 2A: BGB-A333 monotherapy dose expansion (Experimental)
  Interventions: Drug: BGB-A333
- Phase 1B: BGB-A333 and BGB-A317 dose confirmation (Experimental)
  Interventions: Drug: BGB-A333; Drug: BGB-A317
- Phase 2B: BGB-A333 and BGB-A317 dose expansion (Experimental)
  Interventions: Drug: BGB-A333; Drug: BGB-A317

INTERVENTIONS:
Drug: BGB-A333 — Anti-PD-L1 antibody
Drug: BGB-A317 — Anti-PD-1 antibodies
  Other Names: Tislelizumab
  Arms: Phase 1B: BGB-A333 and BGB-A317 dose confirmation; Phase 2B: BGB-A333 and BGB-A317 dose expansion

SUMMARY:
BGB-A333 is a humanized IgG1-variant monoclonal antibody against programmed cell death 1-ligand 1 (PD-L1), the ligand of an immune check point- receptor, programmed cell death-1 (PD-1). BGB-A317 is a humanized, IgG4-variant monoclonal antibody against PD-1. This study tested the safety and anti-tumor effect of BGB-A333 alone and in combination with BGB-A317 in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic disease (unresectable) that is resistant to standard therapy or for which treatment is not available, not tolerated or refused
2. Has Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
3. Has adequate organ function

Key Exclusion Criteria:

1. Active brain or leptomeningeal metastasis.
2. Active autoimmune diseases or history of autoimmune diseases that may relapse.
3. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc. (antiviral therapy is permitted for participants with hepatocellular carcinoma)
4. Concurrent participation in another therapeutic clinical trial.
5. Received prior therapies targeting PD-1 or PD-L1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (8):
- Australia (4):
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Auckland City Hospital, Auckland, New Zealand
- Spain (3):
  - Institut Catala Doncologia, Barcelona
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Desai J, Fong P, Moreno V, Frentzas S, Meniawy T, Markman B, Voskoboynik M, Rahman T, Budha N, Wu J, Marlow J, Yang S, Calvo E, Martin-Liberal J. A Phase 1/2 study of the PD-L1 inhibitor, BGB-A333, alone and in combination with the PD-1 inhibitor, tislelizumab, in patients with advanced solid tumours. Br J Cancer. 2023 Apr;128(8):1418-1428. doi: 10.1038/s41416-022-02128-3. Epub 2023 Feb 16. PMID 36797356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 study centers in Australia, 1 study center in New Zealand, and 3 study centers in Spain. A total of 39 patients were enrolled in the study and all received ≥ 1 dose of study drug.
Groups:
- Phase 1A: BGB-A333 450 mg: BGB-A333 450 mg, intravenously, every 3 weeks
- Phase 1A: BGB-A333 900mg: BGB-A333 900mg, intravenously, every 3 weeks
- Phase 1A: BGB-A333 1350 mg: BGB-A333 1350 mg, intravenously, every 3 weeks
- Phase 1A: BGB-A333 1800 mg: BGB-A333 1800 mg, intravenously, every 3 weeks
- Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg; Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg: BGB-A333 1350 mg, intravenously, + Tislelizumab 200 mg, intravenously, every 3 weeks
Period: Overall Study
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Started | 3 | 3 | 6 | 3 | 12 | 12
Completed | 2 | 2 | 3 | 0 | 3 | 5
Not Completed | 1 | 1 | 3 | 3 | 9 | 7
Not completed — Commenced new anti-cancer therapy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 2 | 1 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 1 | 1 | 4
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Deteriorating condition | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (7.21) | 60.3 (11.24) | 58.8 (14.52) | 58.0 (16.52) | 65.3 (10.85) | 67.5 (8.52) | 63.31 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 2 | 7 | 1 | 18
  Male | 1 | 1 | 2 | 1 | 5 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 6 | 3 | 12 | 11 | 37
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 2 | 12 | 10 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Programmed death-ligand 1 (PD-L1) Status [Number; unit: participants]
  Positive | 0 | 2 | 2 | 1 | 4 | 6 | 15
  Negative | 2 | 1 | 3 | 2 | 7 | 6 | 21
  Missing | 1 | 0 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 and Phase 2 : Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse events were assessed per the National Cancer Institute Common Terminology Criteria for Adverse Events NCI-CTCAE Version 4.03 Serious Adverse Events (SAEs) were monitored from the date of informed consent. All adverse events (AEs) and SAEs, were reported until either 30 days after the last dose of study drug or until initiation of a new anticancer therapy, whichever occurred first.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1A: BGB-A333 900 mg: BGB-A333 900mg, intravenously, every 3 weeks
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12
Participants
  Any Treatment Emergent Adverse Event (TEAE) | 1 | 2 | 6 | 3 | 12 | 12
  Serious TEAE | 0 | 1 | 3 | 1 | 5 | 3

2. Primary Outcome: Phase 1 and Phase 2 : Number of Participants With Abnormalities During Physical Examinations - Ophthalmology Findings
Description: Complete physical examination including an evaluation of 1) head, eyes, ears, nose, throat, 2) cardiovascular, 3) dermatological, 4) musculoskeletal, 5) respiratory, 6) gastrointestinal, and 7) neurological systems was required to be performed at Screening. At subsequent visits (or as clinically indicated), limited, symptom-directed physical examinations were performed. Clinically significant Ophthalmology abnormalities were collected from case report forms. All AEs and SAEs, were reported until either 30 days after the last dose of study drug or until initiation of a new anticancer therapy, whichever occurred first.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1 and Phase 2 : Number of Participants With Abnormal Electrocardiograms (ECG)
Description: Central ECG data was used and the abnormality was determined by the evaluator (Investigating physician). Multiple tests such as QT, HR, PR, RR were used by the evaluator to determine abnormality. All AEs and SAEs, were reported until either 30 days after the last dose of study drug or until initiation of a new anticancer therapy, whichever occurred first.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12
participants | 0 | 1 | 5 | 2 | 1 | 9

4. Primary Outcome: Phase 1 and Phase 2 : Number of Participants With Abnormal Lab Assessment Results
Description: Lab abnormality was based on ANRIND: if the measurement value > upper limit of normal (ULN), it was considered Abnormal. All AEs and SAEs, were reported until either 30 days after the last dose of study drug or until initiation of a new anticancer therapy, whichever occurred first.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12
participants | 3 | 3 | 6 | 3 | 12 | 12

5. Primary Outcome: Phase 1 A: Recommended Phase 2 Dose (RP2D) for BGB-333
Description: RP2D for BGB-A333 alone and in combination with tislelizumab was the maximum tolerated dose (MTD) or less, which was determined by testing increasing doses up to 1800 mg.
Time Frame: Up to 28 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug
Measure: Number; unit: mg
Groups:
- Phase 1A: BGB-A333 Monotherapy Dose Escalation: BGB-A333 450 mg to 1800 mg every three weeks until they were no longer considered to be achieving clinical benefit, showed unacceptable toxicity, or met other discontinuation criteria as determined by the Investigator
Arm/Group | Phase 1A: BGB-A333 Monotherapy Dose Escalation
Number analyzed (Participants) | 15
mg | 1350

6. Primary Outcome: Phase 2B: Overall Response Rate (ORR) Determined by Investigators Based on RECIST Version 1.1
Description: The ORR is defined as the percentage of participants who had confirmed Complete Response (CR) or Partial response (PR) assessed by investigator using RECIST version 1.1
Time Frame: Up to 33.5 months
Population: Safety Analysis Set (also used for efficacy analysis) included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 12
Percentage of participants | 41.7 [15.17 to 72.33]

7. Secondary Outcome: Phase 1A and Phase 1B: Overall Response Rate (ORR) Determined by Investigators Based on RECIST Version 1.1
Description: ORR is defined as the percentage of participants who had confirmed CR or PR assessed by investigator using RECIST version 1.1.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included (also used for efficacy analysis) all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Percentage of participants | 0.0 [0.00 to 70.76] | 33.3 [0.84 to 90.57] | 50.0 [11.81 to 88.19] | 33.3 [0.84 to 90.57] | 16.7 [2.09 to 48.41]

8. Secondary Outcome: Phase 2B: Duration of Response (DOR) Determined by Investigators Based on RECIST Version 1.1
Description: DOR was defined as the time from the first determination of an objective response per RECIST version 1.1, until the first documentation of progression or death, whichever occurs first. DOR was not evaluable in Phase 1A and Phase 1B.
Time Frame: Up to 33.5 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 5
Months | 9.6 [6.0 to NA] — NA = Data not estimable due to insufficient number of participants with events

9. Secondary Outcome: Phase 1 and Phase 2: Disease Control Rate (DCR) Determined by Investigators Based on RECIST Version 1.1
Description: DCR is defined as the percentage of participants with best overall response of CR, PR and Stable Disease.
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12 | 12
Percentage of participants | 33.3 [0.84 to 90.57] | 33.3 [0.84 to 90.57] | 66.7 [22.28 to 95.67] | 66.7 [9.43 to 99.16] | 58.3 [27.67 to 84.83] | 75.0 [42.81 to 94.51]

10. Secondary Outcome: Phase 2B: Progression-free Survival (PFS) Determined by Investigators Based on RECIST Version 1.1
Description: PFS was defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of disease progression assessed by investigator using RECIST v1.1 or death, whichever occurs first
Time Frame: Up to 33.5 months
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 12
Months | 6.1 [1.9 to 11.0]

11. Secondary Outcome: Phase 1: Maximum Plasma Concentration (Cmax) of BGB-A333
Description: PK parameters were derived only for Phase 1A and Phase 1B. Phase 2B pharmacokinetic (PK) parameters were not estimated due to limited sampling.
Time Frame: Cycle 1 Day 1 (Pre-dose, End of infusion, 6 hours), Day 2, Day 4, Day 8, Day 15 and Day 21
Population: The PK analysis population includes all participants with valid PK sampling after treatment with study drug(s)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
μg/mL | 167 (42.4) | 351 (151) | 466 (91.0) | 594 (150) | 455 (127)

12. Secondary Outcome: Phase 1: Time to Cmax (Tmax) of BGB-A333
Description: PK parameters were derived only for Phase 1A and Phase 1B. Phase 2B PK parameters were not estimated due to limited sampling.
Time Frame: Cycle 1 Day 1 (Pre-dose, End of infusion, 6 hours), Day 2, Day 4, Day 8, Day 15 and Day 21
Population: The PK analysis population includes all participants with valid PK sampling after treatment with study drug(s)
Measure: Median (Full Range); unit: Day
Groups:
- Phase 1A: BGB-A333 900 mg: BGB-A333 900 mg, intravenously, every 3 weeks
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Day | 0.05 [0.04 to 0.21] | 0.06 [0.05 to 0.06] | 0.05 [0.05 to 0.22] | 0.06 [0.06 to 0.21] | 0.21 [0.05 to 0.22]

13. Secondary Outcome: Phase 1:Trough Serum Concentration (Ctrough) of BGB-A333
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 (Pre-dose, End of infusion, 6 hours), Day 2, Day 4, Day 8, Day 15 and Day 21
Population: The PK analysis population includes all participants with valid PK sampling after treatment with study drug(s)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
μg/mL | 21.3 (5.69) | 47.0 (26.7) | 90.7 (24.2) | 81.4 (23.9) | 80.0 (22.0)

14. Secondary Outcome: Phase 1: Time to Last Observed Concentration (Tlast) of BGB-A333
Description: PK parameters were derived only for Phase 1A and Phase 1B. Phase 2B PK parameters were not estimated due to limited sampling. Actual observed time values for PK sampling, have an allowable time deviation (+/- 3 days) from the planned nominal time as pre-specified in the Visit Window section of the study protocol.
Time Frame: Cycle 1 Day 1 (Pre-dose, End of infusion, 6 hours), Day 2, Day 4, Day 8, Day 15 and Day 21
Population: The PK analysis population includes all participants with valid PK sampling after treatment with study drug(s)
Measure: Median (Full Range); unit: Day
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 12
Day | 22.0 [21.0 to 22.0] | 21.0 [14.1 to 21.0] | 21.0 [14.0 to 22.0] | 21.0 [21.0 to 24.0] | 21.0 [7.10 to 24.0]

15. Secondary Outcome: Phase 1: Area Under the Concentration-time Curve From 0 to 21 Days Post-dose (AUC 0-21day) of BGB-A333
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 (Pre-dose, End of infusion, 6 hours), Day 2, Day 4, Day 8, Day 15 and Day 21
Population: The PK analysis population includes all participants with valid PK sampling after treatment with study drug(s)
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 2 | 5 | 3 | 11
μg*day/mL | 1095 (141) | 2913 (320) | 3823 (566) | 4141 (648) | 3546 (814)

16. Secondary Outcome: Phase 1A and Phase 2: Number of Participants With Detectable Treatment-Emergent Anti-BGB-A333 Antibodies
Description: Treatment-emergent anti drug antibodies (ADA) was the sum of both treatment-induced ADA and treatment-boosted ADA, synonymous with "ADA Incidence."
Time Frame: Up to 33.5 months
Population: ADA analysis set included participants who received ≥ 1 dose of study drug(s), BGB-A333 in Phase 1A or BGB-A333 and tislelizumab in Phase 1B and Phase 2B and had ≥ 1 evaluable ADA result after treatment.
Measure: Number; unit: participants
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-A333 1350 mg | Phase 1A: BGB-A333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 11 | 12
participants | 1 | 1 | 1 | 0 | 0 | 4

ADVERSE EVENTS:
Time Frame: From the date of consent until study termination (Approximately 33.5 months)
Description: All adverse events were reported until either 30 days after the last dose of study drug or until initiation of a new anticancer therapy, whichever occurred first.
Groups:
- Phase 1A: BGB-A333 450 mg: BGB-333 450 mg, intravenously, every 3 weeks
- Phase 1A: BGB-A333 900 mg: BGB-333 900 mg, intravenously, every 3 weeks
- Phase 1A: BGB-333 1350 mg: BGB-333 1350 mg, intravenously, every 3 weeks
- Phase 1A: BGB-333 1800 mg: BGB-333 1800 mg, intravenously, every 3 weeks
Arm/Group | Phase 1A: BGB-A333 450 mg | Phase 1A: BGB-A333 900 mg | Phase 1A: BGB-333 1350 mg | Phase 1A: BGB-333 1800 mg | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 2/6 | 1/3 | 4/12 | 2/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 3/6 | 1/3 | 5/12 | 3/12
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 6/6 | 3/3 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1A: BGB-A333 450 mg (N=3) | Phase 1A: BGB-A333 900 mg (N=3) | Phase 1A: BGB-333 1350 mg (N=6) | Phase 1A: BGB-333 1800 mg (N=3) | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg (N=12) | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg (N=12)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1A: BGB-A333 450 mg (N=3) | Phase 1A: BGB-A333 900 mg (N=3) | Phase 1A: BGB-333 1350 mg (N=6) | Phase 1A: BGB-333 1800 mg (N=3) | Phase 1B: BGB-A333 1350 mg + Tislelizumab 200 mg (N=12) | Phase 2B (Urothelial Carcinoma Cohort): BGB-A333 1350 mg + Tislelizumab 200 mg (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (7) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 2 (9) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Phase 2A of the study was not initiated nor conducted since BGB-A333 as a monotherapy treatment beyond the completion of dose escalation in Phase 1A was not pursued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03379259/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT03379259/SAP_001.pdf